CLINICAL TRIAL: NCT07068464
Title: Overall Survival Following Interval and Delayed Cytoreduction Surgery in Advanced Stage Ovarian Cancer: a Pragmatic Phase III Randomised Controlled Trial
Brief Title: ICRA Randomised Controlled Trial
Acronym: ICRA
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: NHS Grampian (Other Government)
Responsible Party: Principal Investigator, Faiza Gaba, Dr, University College London Hospitals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: vF_ICRA
Record Dates: First submitted 2025-07-07; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-06

CONDITIONS: Ovary Cancer
Keywords: surgery
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interval cytoreduction surgery (Active Comparator): interval cytoreduction surgery is defined as surgery after 3 cycles of carboplatin and paclitaxel neoadjuvant chemotherapy
  Interventions: Procedure: interval cytoreduction surgery
- delayed cytoreduction surgery (Experimental): delayed cytoreduction surgery is defined as surgery after 6 cycles of carboplatin and paclitaxel neoadjuvant chemotherapy
  Interventions: Procedure: delayed cytoreduction surgery

INTERVENTIONS:
Procedure: delayed cytoreduction surgery — Delayed cytoreduction surgery is defined as cytoreduction surgery after six cycles of carboplatin and paclitaxel neoadjuvant chemotherapy.
  Arms: delayed cytoreduction surgery
Procedure: interval cytoreduction surgery — Interval cytoreduction surgery is defined as cytoreduction surgery after three cycles of carboplatin-paclitaxel neoadjuvant chemotherapy.
  Arms: interval cytoreduction surgery

SUMMARY:
The standard of care for advanced stage epithelial ovarian cancer is primary cytoreduction surgery with the aim of complete cytoreduction, followed by platinum and taxane-based chemotherapy and consideration of maintenance therapy (bevacizumab or Poly ADP-ribose polymerase (PARP)-inhibitor). Neoadjuvant chemotherapy before and after interval cytoreduction surgery has become an alternative approach as randomized controlled trials have demonstrated non-inferiority of this type of management over primary surgery. In these studies, neoadjuvant chemotherapy was restricted to three to four cycles. However, real-world clinical practice varies, with centres giving more than four pre-operative cycles. The decision to delay surgery is complex and influenced by multiple factors. These include poor performance status, radiological evidence of unresectable sites of disease, or insufficient surgical resources (either lack of surgical expertise operating room availability due to waiting lists) particularly when high complexity surgery is required to achieve complete cytoreduction. International disparities in access to surgical resources between high and low-middle income country settings also results in delays to surgery.

Knowledge gap:

There is a paucity of data in the setting of extended use of neoadjuvant chemotherapy (more than four cycles). Data on the role of delayed cytoreduction surgery post four cycles are controversial. While some data have shown survival to be similar to that of patients undergoing interval cytoreductive surgery after three cycles,6-12 others have reported poorer prognosis. Conflicting data are due to selection biases such as heterogeneous inclusion criteria, small sample sizes and retrospective study designs. Delaying surgery to after four cycles has the potential to reduce surgical complexity and post-operative morbidity, and increase rates of complete cytoreduction (an independent marker of survival).

Our multi-centre, international, retrospective cohort study (GO SOAR2) of 2498 women from twenty-two centres across twelve countries with advanced stage ovary cancer, showed that interval cytoreduction surgery was associated with statistically significant greater overall survival in comparison to delayed cytoreduction surgery (HR 0.81, p=0.01) but was associated with a higher GO SOAR surgical complexity score and greater surgical morbidity. Our results indicate that early maximum effort cytoreduction surgery with complete cytoreduction in high volume centres with appropriate surgical skill mix and resources, is what is needed to increase overall survival for women with advanced stage ovarian cancer.

We present the study design for a pragmatic phase III superiority randomised controlled trial comparing overall survival following interval and delayed cytoreductive surgery.

Our hypothesis is that overall survival is greater following interval cytoreduction surgery when compared to delayed cytoreduction in women with stage III-IV epithelial ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Women ≥18 years of age.
2. Histologically confirmed high grade, serous, or endometrioid ovarian cancer, fallopian tube carcinoma, or primary peritoneal carcinoma.
3. International Federation of Gynecologic Oncology (FIGO) 2014 stage IIIA-IVB unsuitable for complete primary cytoreductive surgery because disease unresectable. Assessment of unresectable disease must have been made by staging CT chest abdomen pelvis +/- diagnostic laparoscopy.
4. Disease must be deemed resectable after three courses of neoadjuvant chemotherapy.
5. Patient must be fit for cytoreduction surgery and chemotherapy.

Exclusion Criteria:

1. Women undergoing primary and recurrent cytoreductive surgery.
2. Mucinous, clear cell, carcinosarcoma, low-grade serous carcinoma, germ cell and sex cord stromal histopathologies.
3. Synchronous malignancies.
4. Unfit for surgery and or chemotherapy.
5. Pregnant or breastfeeding women.
6. Delivery of HIPEC at cytoreduction surgery.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 682 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2029-01-31 (Estimated); Study Completion 2034-01-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5 years
  Defined from date of diagnosis to date of death

SECONDARY OUTCOMES:
Progression free survival | 5 years
  Defined from date of diagnosis to date of first recurrence.
Post-operative morbidity | 30 days post surgery
  As per Clavien-Dindo classification.
Peritoneal cancer index (PCI) to assess intra-operative tumour burden and completeness of cytoreduction (CC) | At the end of surgery.
  A measure of extent of residual disease at the end of surgery.
Quality of life as per EQ-5D-5L health-related quality of life questionnaire | 5 years
  Measured using the EQ-5D-5L health-related quality of life questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- University College London Hospitals NHS Foundation Trust, London, United Kingdom